CLINICAL TRIAL: NCT07188441
Title: A Single-center, Single-arm, Open-label Study of the Combination of Teniposide Injection and Cisplatin in the Treatment of Newly Diagnosed Patients With Central Malignant Germ Cell Tumors.
Brief Title: Treatment of Newly Diagnosed Central Malignant Germ Cell Tumor People With Teniposide Injection Combined With Cisplatin.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengcheng Guo (Other)
Responsible Party: Sponsor-Investigator, Chengcheng Guo, MD,Principal Investigator,Clinicial Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNBG-002
Record Dates: First submitted 2024-07-23; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: GCT; Germ Cell Tumor; Central Malignant Germ Cell Tumor
Keywords: Central malignant germ cell tumor; GCT; teniposide; Cisplatin
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Teniposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teniposide plus cisplatin (Experimental): Our study set up only one experimental group without a control group, and all subjects received the same intervention, namely the combination of Teniposide injection and Cisplatin for the treatment of newly diagnosed central malignant germ cell tumor patients. The effectiveness was assessed by observing the results and comparing them with historical data.
  Interventions: Drug: Teniposide Injection

INTERVENTIONS:
Drug: Teniposide Injection — teniposide 300mg/m2 for 5 days, cisplatin 75mg/m2 for 5 days
  Other Names: cisplatin

SUMMARY:
This trial is a prospective single arm intervention study, conducting clinical research on marketed drugs. Adverse drug reactions are controllable and the risk is low, with an estimated total of 40 cases. The main objective is to evaluate the safety and efficacy of teniposide combined with cisplatin in the treatment of newly diagnosed central malignant germ cell tumors, and to conduct drug monitoring on subjects to explore potential biomarkers for predicting therapeutic efficacy. It is expected to ultimately achieve the goal of prolonging the overall survival of patients, while providing more guidance for the screening of the best treatment population and biological predictive markers.

DETAILED DESCRIPTION:
The subjects received an injection of teniposide combined with cisplatin every 3 weeks for one cycle. The teniposide dosage was 300 mg/m2, administered continuously over 3 to 5 days, each time with 500 ml of normal saline through intravenous drip; the cisplatin dosage was 75 mg/m2, also administered continuously over 3 to 5 days, for a total of 4-6 cycles. Radiation therapy was conducted according to standard practices after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Must have at least one measurable lesion defined by RANO criteria
* The initial diagnosis has been confirmed as central malignant germ cell tumor
* Expected survival period ≥ 6 months
* Absolute neutrophil ≥1.0×10^9/L; Platelet ≥100.0×10^9/L
* Aspertate aminotransferase and alanine aminotransferase ≤2.5×Upper limit of normal
* total bilirubin ≤1.5×Upper limit of normal
* Electronic Case Report of Form≥70mL/min/1.73m^2
* Estimated glomerular filtration rate ≥ 70 mL/min/1.73 m² or normal serum creatinine (Cr)
* Women and men with fertility must agree to use appropriate contraceptive methods (hormones or barrier therapy or abstinence) during the study period and within 3 months after the last dose; The pregnancy test of female subjects of childbearing age within 7 days before administration must be negative
* Willing and able to read, understand, and sign written informed consent, parents/guardians of child or adolescent subjects have the ability to understand, agree, and sign research informed consent forms and applicable child consent forms before initiating any protocol related procedures

Exclusion Criteria:

* Patients undergoing any other anti-cancer experimental treatment
* Individuals with a history of severe allergies or allergies to any component of the drugs in the past
* Previous or concurrent active cardiovascular diseases with clinical significance, including congenital heart disease or pericardial disease, history of heart failure, myocardial infarction, coronary heart disease, heart valve disease, cardiomyopathy, and arrhythmia
* Patients with Magnetic Resonance Imaging contraindications
* Those who need to receive live virus vaccine during administration
* Serious complications and/or underlying diseases
* Individuals with poor control of hypertension (under standardized blood pressure reduction protocols, systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 100mmHg)
* Uncontrolled systemic bacterial, viral, or fungal infections
* Patients infected with Human Immunodeficiency Virus(HIV) or syphilis
* Patients who have undergone organ transplantation in the past
* Pregnant or lactating women
* Researchers believe that there are other factors that are not suitable for participating in the experiment

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 3 weeks.
  The proportion of patients who achieved complete response (CR) or partial response (PR) ( i.e. CR PR) from the first use of the investigational drug to the period of withdrawal from the trial, compared to the total number of evaluable cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No